CLINICAL TRIAL: NCT03262467
Title: Aneurysmorrhaphy of Vascular Access for Haemodialysis
Acronym: AVAH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty Hospital Kralovske Vinohrady (Other Government)
Responsible Party: Principal Investigator, Peter Balaz, Principal Investigator, Faculty Hospital Kralovske Vinohrady
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AVAH_V1.0
Record Dates: First submitted 2017-08-23; First posted 2017-08-25 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Patients With an Aneurysm of Native Vascular Access Indicated for Surgical Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aneurysmorrhaphy with external porous prosthesis (Provena©) (Active Comparator)
  Interventions: Procedure: Aneurysmorrhaphy with or without external porous prosthesis (Provena©, BBraun)
- Aneurysmorrhaphy without external porous prosthesis (Placebo Comparator)
  Interventions: Procedure: Aneurysmorrhaphy with or without external porous prosthesis (Provena©, BBraun)

INTERVENTIONS:
Procedure: Aneurysmorrhaphy with or without external porous prosthesis (Provena©, BBraun) — In patients with aneurysm of native vascular access indicated for surgical treatment, aneurysmorrhaphy with or without external porous prosthesis (Provena©, BBraun) wil be performed.

SUMMARY:
In patients with chronic renal failure, a well-functioning vascular access is essential for hemodialysis treatment. Native arteriovenous fistula (AVF) is the first-choice of vascular access, due to a lower incidence of complications and better long-term patency as compared to prosthetic arteriovenous fistula. With the incidence ranging between 6-60%, AVF aneurysm (AAVF) is a common complication of native AVF. According to Kidney Disease Outcomes Quality Initiative (K/DOQI) guidelines, asymptomatic aneurysms are indicated for conservative treatment, but precise recommendations when and how to intervene in available guidelines are missing.

Several surgical (remodeling, resection and substitution, ligation) and endovascular techniques have been described in the AAVF treatment, but there is currently no prospective randomized study comparing these techniques.

In 2008, our team published the first experience with a new surgical method of AAVF treatment - aneurysmorrhaphy with external porous prosthesis (Provena©, BBraun). This therapy was validated in several studies and has shown a good long-term patency and a minimal incidence of complications.

AAVF aneurysmorrhaphy can be performed with or without an external porous prosthesis (Provena©, BBraun). The use of external prostheses reduces venous wall shear stress, turbulent flow, endothelial damage, and thrombus formation, which should improve vascular patency and reduce the risk of AVF re-aneurysm. So far, there is no prospective randomized study comparing the effect of external porous prosthesis on AVF patency and the incidence of postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

1. Signature of informed consent.
2. A male or female subject aged 18 or older.
3. A subject with a naive vascular access aneurysm indicated for surgical treatment.

Exclusion Criteria:

1. Patients with pseudoaneurysm of prosthetic vascular access
2. Patients with a vascular access infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Patency and aneurysms recurrence at 12 months after operation | 12 months

SECONDARY OUTCOMES:
Complications at 12 months | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Faculty Hospital Kralovske Vinohrady, 3rd Medical Faculty, Charles University, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huber TS, Carter JW, Carter RL, Seeger JM. Patency of autogenous and polytetrafluoroethylene upper extremity arteriovenous hemodialysis accesses: a systematic review. J Vasc Surg. 2003 Nov;38(5):1005-11. doi: 10.1016/s0741-5214(03)00426-9. PMID 14603208
- [Background] Salahi H, Fazelzadeh A, Mehdizadeh A, Razmkon A, Malek-Hosseini SA. Complications of arteriovenous fistula in dialysis patients. Transplant Proc. 2006 Jun;38(5):1261-4. doi: 10.1016/j.transproceed.2006.02.066. PMID 16797276
- [Background] Sidawy AN, Spergel LM, Besarab A, Allon M, Jennings WC, Padberg FT Jr, Murad MH, Montori VM, O'Hare AM, Calligaro KD, Macsata RA, Lumsden AB, Ascher E; Society for Vascular Surgery. The Society for Vascular Surgery: clinical practice guidelines for the surgical placement and maintenance of arteriovenous hemodialysis access. J Vasc Surg. 2008 Nov;48(5 Suppl):2S-25S. doi: 10.1016/j.jvs.2008.08.042. PMID 19000589
- [Background] Balaz P, Rokosny S, Klein D, Adamec M. Aneurysmorrhaphy is an easy technique for arteriovenous fistula salvage. J Vasc Access. 2008 Apr-Jun;9(2):81-4. PMID 18609522
- [Background] Berard X, Brizzi V, Mayeux S, Sassoust G, Biscay D, Ducasse E, Bordenave L, Corpataux JM, Midy D. Salvage treatment for venous aneurysm complicating vascular access arteriovenous fistula: use of an exoprosthesis to reinforce the vein after aneurysmorrhaphy. Eur J Vasc Endovasc Surg. 2010 Jul;40(1):100-6. doi: 10.1016/j.ejvs.2010.01.021. Epub 2010 Mar 3. PMID 20202869
- [Background] Rokosny S, Balaz P, Wohlfahrt P, Palous D, Janousek L. Reinforced aneurysmorrhaphy for true aneurysmal haemodialysis vascular access. Eur J Vasc Endovasc Surg. 2014 Apr;47(4):444-50. doi: 10.1016/j.ejvs.2014.01.010. Epub 2014 Jan 21. PMID 24530180
- [Background] Wohlfahrt P, Rokosny S, Melenovsky V, Borlaug BA, Pecenkova V, Balaz P. Cardiac remodeling after reduction of high-flow arteriovenous fistulas in end-stage renal disease. Hypertens Res. 2016 Sep;39(9):654-9. doi: 10.1038/hr.2016.50. Epub 2016 May 26. PMID 27225601
- [Background] Barra JA, Volant A, Leroy JP, Braesco J, Airiau J, Boschat J, Blanc JJ, Penther P. Constrictive perivenous mesh prosthesis for preservation of vein integrity. Experimental results and application for coronary bypass grafting. J Thorac Cardiovasc Surg. 1986 Sep;92(3 Pt 1):330-6. PMID 3528676
- [Background] Meguro T, Nakashima H, Kawada S, Tokunaga K, Ohmoto T. Effect of external stenting and systemic hypertension on intimal hyperplasia in rat vein grafts. Neurosurgery. 2000 Apr;46(4):963-9; discussion 969-70. doi: 10.1097/00006123-200004000-00036. PMID 10764272